CLINICAL TRIAL: NCT03821909
Title: Acquisition of Portal Venous Circulating Tumor Cells and Exosomes From Patients With Pancreatic Cancer by Endoscopic Ultrasound: a Prospective Study
Brief Title: Acquisition of Portal Venous CTCs and Exosomes From Patients With Pancreatic Cancer by EUS
Acronym: CTCs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ying Lv (Other)
Responsible Party: Sponsor-Investigator, Ying Lv, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Other Study IDs: EPCE-1
Record Dates: First submitted 2019-01-06; First posted 2019-01-30 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Portal venous blood; Circulating tumor cells; Exosome
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will obtain portal venous blood samples via endoscopic ultrasound(EUS) in patients with suspected pancreatic masses, detect circulating tumor cells and analyze the mRNA markers of the exosomes by RNA-seq.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreatic cancer: Endoscopic ultrasound-guided protal venous blood sampling will be performed for each patient. And the diagnosis will be confirmed by tissue pathology.
  Interventions: Procedure: Endoscopic ultrasound-guided protal venous blood sampling
- Benign pancreatic diseases: Endoscopic ultrasound-guided protal venous blood sampling will be performed for each patient. And the diagnosis will be confirmed by tissue pathology, e.g. PCLs.
  Interventions: Procedure: Endoscopic ultrasound-guided protal venous blood sampling

INTERVENTIONS:
Procedure: Endoscopic ultrasound-guided protal venous blood sampling — We wil obtain portal venous blood samples via endoscopic ultrasound(EUS) in patients with suspected pancreatic masses.

SUMMARY:
The investigators are going to explore the diagnostic and prognostic value of circulating tumor cells and exosomes extracted from the portal venous blood obtained with endoscopic ultrasound in pancreatic cancer patients.

DETAILED DESCRIPTION:
As the prognosis of pancreatic cancer, a kind of malignant tumor, remains poor due to the low diagnostic rate at the early stage, there is still a significant clinical need to determine individualized tumor molecular profiles and personalized risk for recurrence. Circulating tumor cells (CTCs) and exosomes from patients with primary tumors may hold promise in serving as an informative biomarker to address this clinical need. Here in this study, the investigators are going to explore the feasibility and safety of sampling portal venous blood via endoscopic ultrasound (EUS), and detect portal venous CTCs and analyze mRNA markers of exosomes by RNA-seq. The investigators aim to explore the potential molecular mechanisms in tumor microenvironment and mechanisms of drug resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 80 years-old
2. Suspected pancreatic masses and referred for EUS-FNA for pathology diagnosis
3. Written informed consent

Exclusion Criteria:

1. Patients who have received adjuvant chemotherapy and other anti-tumor treatments
2. Severe heart, lung, liver, kidney insufficiency, or severe bleeding disorders, severe coagulopathy or local/systemic infections, other critical illnesses
3. Women who are planning to become pregnant or are pregnant or breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suspected to have pancreatic masses who are going to receive EUS-FNA operations for diagnostic purposes.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
The difference of the amount of circulating tumor cells acquisited from portal venous blood between patients with pancreatic cancer and benign pancreatic diseases | 08/01/2018-08/01/2020
  In this study, the amount of the circulating tumor cells obtained from portal venous blood of suspected pancreatic masses patients will be determined by analyzing the expression of folate receptors. The investigators will compare the difference of the CTC amount between patients with pancreatic cancer and benign pancreatic diseases.
The difference of the exosomes acquisited from portal venous blood between patients with pancreatic cancer and benign pancreatic diseases | 08/01/2018-08/01/2020
  Exosomes will be acquisited from portal venous blood of patients with suspected pancreatic masses. Then the total RNA will be extracted from the exosomes. The investigators will compare the expression of certain mRNA markers of the exosomes between patients with pancreatic cancer and benign pancreatic diseases. (The mRNA markers will be selected from RNA-seq results.)

SECONDARY OUTCOMES:
The difference of the amount of circulating tumor cells between portal venous and peripheral blood | 08/01/2018-08/01/2020
  In this study, the amount of the circulating tumor cells obtained from portal venous blood and peripheral blood will be assessed for each patient respectively. The investigators will compare the difference of the CTC amount between portal venous blood and peripheral blood.
The difference of the exosomes between portal venous and peripheral blood | 08/01/2018-08/01/2020
  Exosomes will be acquisited from portal venous blood and peripheral blood for each patient. Then the total RNA will be extracted from the exosomes. The investigators will compare the expression of certain mRNA markers of the exosomes between portal venous and peripheral blood for each patient. (The mRNA markers will be selected from RNA-seq results.)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lv, PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided